CLINICAL TRIAL: NCT06370013
Title: An Open Label, Multicenter Rollover Study for Continued Characterization of Safety and Tolerability of TT-00420 (Tinengotinib) Tablet Monotherapy in Adult Patients With Advanced Solid Tumors
Brief Title: Rollover Study to Provide Continued Access to TT-00420 (Tinengotinib) for Subjects With Advanced Solid Tumors
Status: Available | Type: Expanded Access
Sponsor: TransThera Sciences (Nanjing), Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TT00420US14
Record Dates: First submitted 2024-04-09; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Advanced Solid Tumors; Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Tinengotinib — Subjects on this rollover study may continue to receive tinengotinib at the dose that they were previously receiving on the TransThera parent study. Dose may be decreased by one dose level from the previously-received dose upon study entry, based on physician discretion.
  Other Names: TT-00420

SUMMARY:
This study is an open-label, multicenter study for Continued Characterization of Safety and Tolerability of TT-00420 (tinengotinib) Tablet Monotherapy in Adult Patients with Advanced Solid Tumors

DETAILED DESCRIPTION:
This is a Rollover study. Only subjects who continue to receive clinical benefit from continuation of tinengotinib monotherapy and are tolerating tinengotinib at the time of enrollment are eligible to participate on this study. Subjects on this rollover study may continue to receive tinengotinib at the dose that they were previously receiving on the TransThera parent study and may continue for as long as the subject continues to benefit from treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is currently enrolled in a pre-defined TransThera-sponsored parent study and is receiving tinengotinib as a single agent.
2. Subject is currently deriving clinical benefit from the study treatment, as determined by the investigator.

Exclusion Criteria:

1. Subject has been permanently discontinued from tinengotinib in the parent protocol for any reason other than enrollment in the Rollover study
2. Subject does not meet the criteria specified in the parent protocol for continued treatment on study.

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of Chicago Medical Center, Chicago, Illinois
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - UW Carbone Cancer Center, Madison, Wisconsin